CLINICAL TRIAL: NCT06585098
Title: The Effect of Game-Based Virtual Reality Application on the Development of Postoperative Care Skills of Nursing Students for Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, ELMAS DÖNMEZ, principal investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EGE-SBE-KSHA-EMD-01
Record Dates: First submitted 2024-07-18; First posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nursing; Hysterectomy; Game-Based Learning

STUDY DESIGN:
Intervention Model Description: The intervention is a study with an experimental model with a control group.
Who Masked: Participant
Masking Description: The study was planned with two groups (control, intervention). In order to prevent information sharing between groups, at the beginning of the research, the students involved in the study were asked to keep the information and documents given to them confidential. In addition, in order to prevent influence and information exchange, the control group was first invited to the application, then the game was sent to the intervention group and they were allowed to play the game for a week, and then the intervention group was put into the application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group experienced game-based virtual reality application in addition to standard training and hybrid simulation.
  Interventions: Other: game based learning
- control group (No Intervention): The control group experienced standard training and hybrid simulation

INTERVENTIONS:
Other: game based learning — The students in the intervention group were informed by the researcher, and the students who met the research participation criteria and volunteered to participate in the research filled out the "Informed Consent Form (Annex 1)" and downloaded the prepared game-based virtual reality application by entering the prepared website and using their username and password for a period of 1 week. They were asked to play with. After one week, students in the intervention group were invited to a simulation-based training application in groups of seven. In addition, the game was played at least once by the students in the intervention group under the supervision of the researcher.
  Arms: intervention group

SUMMARY:
This study aimed to determine the effect of game-based virtual reality application on nursing students' self-confidence in postoperative care knowledge, skills, satisfaction and learning following hysterectomy surgery.

DETAILED DESCRIPTION:
Method: A total of 179 third-year students studying in the third year of Ege University Faculty of Nursing in the fall semester of 2023-2024 were included in this study, who had the theoretical knowledge about Gynecology and Obstetrics Nursing within the scope of the Diseases and Nursing Care II course, were in the practice of Gynecology and Obstetrics Nursing, and voluntarily agreed to participate in the study. The students were divided into two groups, 42 control and 42 intervention groups, using simple random sampling method. Prior written consent was obtained from both the ethics committee and the institution for conducting the study. Data collection instruments included a Demographic Data Collection Form, a Form for Determining Student Opinions Regarding Game-Based Virtual Reality Application, a Postoperative Care Knowledge Test for Hysterectomy Surgery, a Satisfaction with Education Methods Questionnaire, and the Student Satisfaction and Confidence in Learning Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 3rd year internship of Women's Health and Diseases Nursing Course,
* Having internet access,
* Being able to use a computer,
* Volunteering to participate in the research.

Exclusion Criteria:

* Being a graduate of Health Vocational High School,
* Working as a nurse,
* Taking the Women's Health and Diseases Nursing Course 3rd year internship for the second time

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Educational Methods Survey | immediately after game-based virtual reality application and simulation method
  This is a survey developed by Gürpınar and also used in his research. This survey consists of 16 statements. One of these statements is the statement that asks whether or not the student is satisfied with the education by saying "I am generally satisfied with this educational method". The other statements are generally composed of statements that can determine the opinions about the effect of the educational method on learning and future working life. It is prepared in a 5-Likert type and is scored from 1- strongly disagree to 5- strongly agree, as the score increases, the satisfaction with the educational method is measured and as the score decreases, the dissatisfaction with the method is measured. A minimum of 16 and a maximum of 80 points can be obtained in the evaluation.
Student Satisfaction and Self-Confidence in Learning Scale | immediately after simulation method
  The scale has two sub-dimensions and 13 statements presented as "satisfaction with learning" and "self-confidence". The expressions of satisfaction with learning; "comfort with the learning system", "variety of learning rates", "facilitation", "motivation" and five statements evaluating the suitability of the simulation, the expressions of self-confidence; "adequacy in scope", "necessity of content", "skill improvement", "available resources" and information on how to get help to solve clinical problems in the simulation. It was coded as the 13th item in the scale. A 5-point Likert type was prepared and 1-definitely disagree and 5-definitely complete until the score is given. The minimum score that can be obtained is 13, the maximum score is 65. It is understood that happiness and self-confidence increase as the score increases. The internal discounts of the scale change as 0.94.
Postoperative Care Knowledge Test After Hysterectomy Surgery | immediately before and after simulation application
  This test was created by the researcher in accordance with the relevant literature in order to determine the knowledge levels of students regarding postoperative care after total abdominal hysterectomy surgery.The test consists of 11 questions, 1 point is calculated for each question answered correctly, and the highest score is prepared according to the number of questions. The prepared knowledge test was evaluated by five experts specialized in Women's Health and Diseases Nursing and their suggestions were received. The necessary changes were made to the knowledge test with the suggestions received and its final form was given.
Management of Postoperative Care After Hysterectomy Surgery Clinical Skills Guide | during simulation application
  This is a clinical skill guide created by the researcher in accordance with the relevant literature. "Management of Postoperative Care After Hysterectomy Surgery Clinical Skills Guide" was created to measure the procedures that students will perform in the hybrid simulation application and to benefit from the meeting to be held with educators and students after the application. The statements were scored from 1 to 3 and prepared in the form of a 3-point Likert scale.Maximum 45, minimum 15 points can be obtained and the high score obtained shows the competence of the students. Opinions were received from 8 experts regarding the ''Clinical Skills Guide for Management of Postoperative Care After Hysterectomy Surgery''. Expert opinion analysis was performed and the Content Validity Index (CVI) was found to be 0.944.
Form for Determining Students' Opinions on Game-Based Virtual Reality Application | immediately after the game-based virtual reality application
  This form was developed by the researcher by reading the relevant literature to determine whether students were satisfied or not based on their evaluations regarding the teaching of postoperative care after hysterectomy using a game-based virtual reality application. The form consists of 16 propositions. Students chose one of the three-point Likert-type statements (agree, partially agree, disagree).

CONTACTS AND LOCATIONS:
Locations (1):
- Ege Üniversitesi Kadın Sağlığı Ve Hemşireliği, Izmir, Eyalet/Yerleşke, Turkey (Türkiye)